CLINICAL TRIAL: NCT00318188
Title: Effects of a Personalized Standardized Rehabilitation Program on the Quality of Life of Patients With Systemic Sclerosis Patients : a Randomized Controlled Trial
Brief Title: Effects of a Personalized Standardized Rehabilitation Program in Systemic Sclerosis
Acronym: SCLEREDUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AOM04023
Record Dates: First submitted 2006-04-25; First posted 2006-04-26 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Systemic Scleroderma
Keywords: scleroderma; HAQ; Intensive care reeducation, readaptation
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The patients in this group will do a personalized standardized rehabilitation program on the quality of life.
  Interventions: Procedure: standardized reeducation and readaptation program
- Control group (No Intervention): Habitual care

INTERVENTIONS:
Procedure: standardized reeducation and readaptation program
  Arms: Intervention group

SUMMARY:
Systemic sclerosis (SSc) is a connective-tissue disease characterized by excessive collagen deposition, vascular hyper-reactivity and obliterative microvascular phenomena leading to disability, handicap, and worsening of quality of life. Pharmacological treatments are mainly used for vascular involvement. To date, no pharmacological treatment have been shown to be effective for the fibrosis leading to skin, tendon, and joint disability. Our hypothesis is that rehabilitation could be an interesting non pharmacological treatment in order to decrease the handicap of SSc patients. Our objective is to evaluate the effect of a personalized standardized rehabilitation program on the quality of life of SSc patients in a multicentric randomized controlled trial. This trial will compare a personalized standardized rehabilitation program to the usual non pharmacological treatment. The primary outcome measure will be the HAQ DI (Health Assessment Questionnaire Disability Index). A Zelen design will be used for this study.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged from 18 years or more, with diagnostic of SSc considering the ACR and/or Leroy and Medsger's criteria.
* HAQ greater than or equal to 0.5
* A perception of limitation of mouth opening and/or at least one limitation in range of motion due to illness
* Good understanding of the French language

Exclusion Criteria :

* Associated chronic handicap diseases (stroke, multiple sclerosis, amyotrophic lateral sclerosis, Parkinson's disease, amputated ....)
* Any underlying disease that may be incompatible with the management, discovery at the inclusion visit
* Cognitive problems making it impossible to assess the primary outcome measure
* Patients with a standardized rehabilitation program within 6 months prior to inclusion
* Impairment of comprehension or expression of the French language
* Patients participating in another clinical trial or participated in another clinical trial in the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
HAQ DI:Health Assessment questionnaire disability index | at 12 months
  Health Assessment questionnaire disability index

SECONDARY OUTCOMES:
Mac Tar (Mc Master Toronto Arthritis questionnaire) | at 12 months
  Mc Master Toronto Arthritis questionnaire
S-HAQ ( scleroderma-modified health assessment questionnaire) | at 12 months
  Scleroderma-modified health assessment questionnaire
SF 36 | at 12 months
Kapandji modified index | at 12 months
Rodnan score | at 12 months
Hand Cochin Function Scale | at 12 months
Pain | at 12 months
Mouth opening | at 12 months
Forced expiratory volume (FEV) | at 12 months
Satisfaction of clinical condition | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Serge POIRAUDEAU, MD-PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Reeducation and readaptation Department, Paris, France

REFERENCES:
- [Result] Papelard A, Daste C, Alami S, Sanchez K, Roren A, Segretin F, Lefevre-Colau MM, Rannou F, Mouthon L, Poiraudeau S, Nguyen C. Construction of an ICF core set and ICF-based questionnaire assessing activities and participation in patients with systemic sclerosis. Rheumatology (Oxford). 2019 Dec 1;58(12):2260-2272. doi: 10.1093/rheumatology/kez209. PMID 31219594
- [Result] Rannou F, Boutron I, Mouthon L, Sanchez K, Tiffreau V, Hachulla E, Thoumie P, Cabane J, Chatelus E, Sibilia J, Roren A, Berezne A, Baron G, Porcher R, Guillevin L, Ravaud P, Poiraudeau S. Personalized Physical Therapy Versus Usual Care for Patients With Systemic Sclerosis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2017 Jul;69(7):1050-1059. doi: 10.1002/acr.23098. Epub 2017 Jun 7. PMID 27696703
- [Derived] Daste C, Rannou F, Mouthon L, Sanchez K, Roren A, Tiffreau V, Hachulla E, Thoumie P, Cabane J, Chatelus E, Sibilia J, Poiraudeau S, Nguyen C. Patient acceptable symptom state and minimal clinically important difference for patient-reported outcomes in systemic sclerosis: A secondary analysis of a randomized controlled trial comparing personalized physical therapy to usual care. Semin Arthritis Rheum. 2019 Feb;48(4):694-700. doi: 10.1016/j.semarthrit.2018.03.013. Epub 2018 Mar 27. PMID 29685482